CLINICAL TRIAL: NCT05244889
Title: Digital Cognitive Behaviour Therapy for Insomnia in Chronic Migraines: Feasibility of a Randomised Controlled Trial
Brief Title: Digital CBTI for Comorbid Insomnia in Chronic Migraine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Strathclyde (Other)
Responsible Party: Principal Investigator, Megan Crawford, Principal Investigator, University of Strathclyde
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRUK 202021-29
Record Dates: First submitted 2021-07-07; First posted 2022-02-17 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Insomnia Chronic; Migraine Disorders
Keywords: Cognitive Behaviour Therapy; Digital Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned to a dCBT-I or the sleep hygiene education control group.
Who Masked: Outcomes Assessor
Masking Description: While the study will be single-blinded (researchers analysing data will be blind to allocation), randomisation will be concealed to the RA and participant until the individual's eligibility has been established.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital CBT-I (Experimental): After assignment to dCBT-I, participants will complete a baseline assessment of their sleep, migraines and other outcomes and complete a 30-day sleep and headache diary, and wear an actigraphy device for 7 days to record their sleep and light exposure. They will then be given access to the 6-session dCBT-I programme. At month 1, participants will wear an actigraph device for 1 week.. At month 3 participants will complete a 30-day post-treatment assessment including a sleep and headache diary and the same battery of questionnaires as during the baseline assessment. A subset of participants (and providers) will be invited to participate in an interview about uptake of dCBT-I. At month 6, all participants will complete follow-up questionnaires (similar to baseline and post-treatment questionnaires) and one last 30-day assessment of sleep and headaches and wear a 7-day actigraphy device.
  Interventions: Behavioral: Digital CBT-I
- Sleep Hygiene Education (SHE) (Active Comparator): After assignment to SHE, participants will complete a baseline assessment of their sleep, migraines and other outcomes and complete a 30-day sleep and headache diary, and wear an actigraphy device for 7 days to record their sleep and light exposure. They will then be given access to the 6-session SHE programme. At month 1, participants will wear an actigraph device for 1 week.. At month 3 participants will complete a 30-day post-treatment assessment including a sleep and headache diary and the same battery of questionnaires as during the baseline assessment. A subset of participants (and providers) will be invited to participate in an interview about uptake of SHE. At month 6, all participants will complete follow-up questionnaires (similar to baseline and post-treatment questionnaires) and one last 30-day assessment of sleep and headaches and wear a 7-day actigraphy device.
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: Digital CBT-I — The digital CBT-I intervention (www.sleepio.com) consists of six weekly sessions of CBT-I delivered over the internet by an animated virtual therapist known as "The Prof". The content includes behavioral (e.g. sleep restriction, stimulus control), cognitive (e.g. putting the day to rest, thought re-structuring, mindfulness) strategies, relaxation strategies (e.g., progressive muscle relaxation) and advice on lifestyle and bedroom factors (sleep hygiene). Although the sessions can be completed at the persons own pace, the shortest interval between individual sessions is 7 days, thus participants can complete the course in 6 weeks, or take as long as 12 weeks. As part of the SLEEPIO program, participants will be required to enter their sleep/wake patterns using electronic sleep diaries. There is no face-to-face contact throughout the intervention and all treatment sessions, support and reminders are provided through the online platform.
  Arms: Digital CBT-I
Behavioral: Sleep Hygiene Education — Sleep Hygiene Education (SHE) has successfully been used as a control condition in other trials evaluating dCBT-I42. SHE does not have any therapeutic benefits for individuals with insomnia alone, but is often part of usual care. Consequently it is a credible alternative to dCBT-I. The sleep hygiene education will be provided on a website with access to information about lifestyle changes (e.g., reducing exercise in the evening, light snack before bedtime, reducing caffeine) and changes to the bedroom environment (e.g., dark room, comfortable mattress, optimal room temperature). As with the dCBT-I group, participants will not be required to make any changes to their usual care.
  Arms: Sleep Hygiene Education (SHE)

SUMMARY:
The overall aims of the study are:

Aim 1: Estimate effect sizes: To estimate the effects of dCBT-I on insomnia symptoms compared to a control group (sleep hygiene education) and estimate the relationship between changes in insomnia symptoms and the reduction in migraines.

Aim 2: Explore mechanisms of change: To explore the mechanisms underlining the change in migraine symptoms.

Aim 3: Assess barriers to conducting a full-scale RCT: To collect data on recruitment pace and dropouts in both groups, which will help refine the methodology and maximise uptake and retention of a full-scale randomised control trial (RCT). The investigators will conduct qualitative interviews with a select number of participants and practitioners to identify motivators/barriers in uptake of a digitalised version of CBT-I.

DETAILED DESCRIPTION:
Chronic migraine (CM) is a debilitating condition that places a direct burden worth £150 million on the NHS per year. Previous research has shown that insomnia is a risk factor for migraines. The investigators hypothesise that two modifiable behaviours explain this relationship between insomnia and migraines: daytime napping and nocturnal light exposure. To cope with the migraines, individuals will nap during the day, reducing the homeostatic drive for sleep at night and delaying sleep onset. This inability to fall asleep potentially increases exposure to evening bright light, delaying the release of the hormone melatonin and reducing sleep quality. Poor sleep in turn is a trigger for migraines, which creates a vicious cycle of migraines and poor sleep. The investigators believe that these behavioural mechanisms are valid targets for treatment and are explicitly addressed in Cognitive Behaviour Therapy for insomnia (CBT-I). Digital versions of CBT-I (dCBT-I) offer a scalable solution to the problem of limited access to CBT-I. This research group has demonstrated the feasibility, acceptability and preliminary efficacy of dCBT-I in an uncontrolled proof-of concept study. Utilising randomised control trial (RCT) methodology, the investigator's aim now is to evaluate the effectiveness of dCBT-I for improving insomnia and migraines in patients with chronic migraines. The second aim is to probe mechanism of change and to test the hypotheses that behavioural markers such as daytime napping and evening light exposure can reduce insomnia symptoms leading to an improvement in migraines. Prior to progressing to a full-scale RCT, the investigators require a feasibility RCT, to refine the methodology. The investigators propose to recruit individuals who meet criteria for CM and insomnia, directly referred from two neurology clinics, who will act as clinical recruiters. Eighty-eight participants will be randomised either to a dCBT-I group or to sleep hygiene education (SHE) control group. The main outcomes are insomnia and migraine days and will be collected at post-treatment, and long-term effects will be assessed at month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18 and above
2. Insomnia, satisfied by a total score ≥ 11 on the insomnia severity index (ISI)
3. Headache ≥ 15 days per month, ≥ 12 months and meet criteria for migraine with/without aura on ≥ 8 days per month, ≥ 12 months

Exclusion Criteria:

1. Medical condition that is unstable, requires immediate treatment, or is judged to interfere with the protocol, including other pain conditions such as chronic low back pain and fibromyalgia and also sleep disorders such as untreated sleep apnoea or parasomnias.
2. Psychiatric condition that is judged to interfere with the study protocol including substance abuse, psychotic disorder, cognitive disorder, current suicidal ideation, or any uncontrolled psychiatric conditions that require immediate treatment
3. Regular use of illegal substances
4. Women who are pregnant or breastfeeding
5. Shiftworkers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity | Posttreatment (3 months after intervention starts).
  The change in insomnia (measured with the Insomnia Severity Index - ISI) from baseline to posttreatment. The ISI is scored from 0 to 28, where a higher score indicates more severe insomnia severity.
Change in Migraine Days | Posttreatment (3 months after intervention starts).
  The change in migraine days (measured with the headache diary) from baseline to posttreatment
Recruitment rate | Monthly throughout study completion
  How many participants have been recruited per month
Retention rate | Through study completion, up to 3 years
  How many participants have dropped out
Naps | Mid treatment (Month 1-2 of study)
  Number (N) of naps
Light exposure | Mid treatment (Month 1-2 of study)
  Light exposure measured through an actigraphy device
Barriers and Facilitators to Engagement with the protocol | Post-treatment (3 months after the intervention started)
  Measured through qualitative interviews/focus groups

SECONDARY OUTCOMES:
Adverse Events | Through study completion, up to 3 years
  Adverse Events
Treatment Satisfaction | Post-treatment (3 months after the intervention started)
  Measured through in house post-treatment satisfaction questionnaire
Migraine Disability | Post-treatment (3 months after the intervention started)
  Measured with Migraine Disability Assessment (MIDAS) questionnaire
Medication use | Post-treatment (3 months after the intervention started)
  Captured through headache diaries
Depression and Anxiety | Post-treatment (3 months after the intervention started)
  Captured with the Four-Item Patient Health Questionnaire (PHQ-4) for Anxiety and Depression
Cost-utility | Post-treatment (3 months after the intervention started)
  Measured with the EQ-5D, health-related quality of life, from which quality adjusted life years (QUALY) can be obtained. This will allow us to calculate cost-utility.
Sleepiness | Post-treatment (3 months after the intervention started)
  Measured with Epworth Sleepiness Scale
Fatigue | Post-treatment (3 months after the intervention started)
  Measured with Flinders Fatigue Scale (FFS)

CONTACTS AND LOCATIONS:
Overall Officials: Louise McKean, Study Chair — University of Strathclyde
Locations (2):
- United Kingdom (2):
  - Glasgow, Glasgow
  - Walton Centre, Liverpool, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code